CLINICAL TRIAL: NCT03990571
Title: A Phase 2 Clinical Trial of Axitinib and Avelumab in Patients With Recurrent/Metastatic Adenoid Cystic Carcinoma (ACC)
Brief Title: Axitinib and Avelumab in Treating Patients With Recurrent or Metastatic Adenoid Cystic Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0107; NCI-2019-03704 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0107 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Results first posted 2024-08-26 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Adenoid Cystic Carcinoma; Progressive Disease; Recurrent Adenoid Cystic Carcinoma
MeSH Terms: conditions — Carcinoma, Adenoid Cystic; Disease Progression | interventions — avelumab; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (axitinib, avelumab) (Experimental): Patients receive axitinib PO BID on days 1-28 and avelumab IV over 1 hour on days 1 and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Avelumab; Drug: Axitinib

INTERVENTIONS:
Drug: Avelumab — Given IV
  Other Names: Bavencio; MSB-0010718C; MSB0010718C
Drug: Axitinib — Given PO
  Other Names: AG-013736; AG013736; Inlyta

SUMMARY:
This phase II trial studies how well axitinib and avelumab work in treating patients with adenoid cystic carcinoma that has come back or spread to other places in the body. Axitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as avelumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving axitinib and avelumab together may help to control adenoid cystic carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the objective response rate (ORR) to axitinib and avelumab combination according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria patients with recurrent or metastatic adenoid cystic carcinoma (ACC) who have evidence of disease progression within 6 months prior to study enrollment.

SECONDARY OBJECTIVES:

I. Assess ORR to axitinib and avelumab combination according to immune-related (ir)RECIST criteria patients with recurrent or metastatic adenoid cystic carcinoma (ACC).

II. Evaluate median progression free survival (PFS), PFS rate at 6 months after start of treatment.

III. Evaluate median overall survival (OS), OS rate at 6 months after start of treatment.

IV. Evaluate duration of response (DoR). V. Evaluate safety and toxicity.

EXPLORATORY OBJECTIVES:

I. Assess molecular markers associated with response and resistance to the study combination using tissue and/or plasma obtained from study participants.

OUTLINE:

Patients receive axitinib orally (PO) twice daily (BID) on days 1-28 and avelumab intravenously (IV) over 1 hour on days 1 and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 and 90 days and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group ECOG performance status 0 or 1
* Histologically confirmed recurrent or metastatic adenoid cystic carcinoma not amenable to curative intent surgery or radiotherapy
* Measurable disease per RECIST 1.1
* Evidence of disease progression within 6 months of study enrollment or worsening disease-related symptoms
* Previously untreated subjects and subject treated with any number of prior lines of therapy are eligible
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelet count >= 100 x 10^9/L
* Hemoglobin >= 9 g/dL (may have been transfused)
* Total bilirubin level =< 1.5 x the upper limit of normal (ULN) range
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels =< 2.5 x ULN or AST and ALT levels =< 5 x ULN (for subjects with documented metastatic disease to the liver)
* Estimated creatinine clearance >= 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method)
* Must have archival tissue (formalin-fixed, paraffin-embedded [FFPE] tissue available-minimum of 15 unstained slides) or be willing to undergo a biopsy
* For patients receiving anti-therapeutic coagulation, patients must be on stable anticoagulant regimen and international normalized ratio (INR) or activated partial thromboplastin time (aPTT) must be =< 1.5 upper limit of normal
* Females of childbearing potential must not be breast feeding and must have a negative serum or urine pregnancy test and must agree to use highly effective contraception for a minimum of two weeks prior to receiving study medication until 30 days after discontinuation of the study medication. Acceptable methods of contraception include total and true sexual abstinence, hormonal contraceptives that are not prone to drug-drug interactions (intra uterine system [IUS] levonorgestrel intra uterine system [Mirena], medroxyprogesterone injections [Depo-Provera]), copper-banded intra-uterine devices, and vasectomized partner. All hormonal methods of contraception should be used in combination with the use of a condom by their sexual male partner. Females of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause)
* Women will be considered post-menopausal if they have been amenorrheic for the past 12 months without an alternative medical cause. The following age-specific requirements must also apply: Women < 50 years old: they would be considered post-menopausal if they have been amenorrheic for the past 12 months or more following cessation of exogenous hormonal treatments. The levels of luteinizing hormone (LH) and follicle-stimulating Hormone (FSH) must also be in the post menopausal range (as per the institution). Women >= 50 years old: they would be considered post-menopausal if they have been amenorrheic for the past 12 months or more following cessation of all exogenous hormonal treatments, or have had radiation-induced oophorectomy with the last menses > 1 year ago, or have had chemotherapy-induced menopause with > 1 year interval since last menses, or have had surgical sterilization by either bilateral oophorectomy or hysterectomy
* Non-sterilized males who are sexually active with a female partner of childbearing potential must use adequate contraception for the duration of the study and 30 days after the last dose of study medication. Adequate contraception methods include: birth control pills (e.g. combined oral contraceptive pill), barrier protection (e.g. condom plus spermicide, cervical/vault cap or intrauterine device), and abstinence. Patients should not father a child for 6 months after completion of the study medication. Patients should refrain from donating sperm from the start of dosing until 6 months after discontinuing the study medication. If male patients wish to father children they should be advised to arrange for freezing of sperm samples prior to the start of the study medication
* For patients with hypertension, upon entry into study must have blood pressure of < 140/90
* Corrected QT interval (QTc) < 470 msec

Exclusion Criteria:

* Current use of immunosuppressive medication, EXCEPT for the following:

  * Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection)
  * Systemic corticosteroids at physiologic doses =< 10 mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication)
* Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible
* Prior organ transplantation including allogenic stem-cell transplantation
* Active infection requiring systemic therapy
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome
* Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV ribonucleic acid [RNA] if anti-HCV antibody screening test positive)
* Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version [v]4.03 grade >= 3)
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (>= New York Heart Association Classification class II), or serious cardiac arrhythmia requiring medication
* Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 grade > 1); however, alopecia, sensory neuropathy grade =< 2, or other grade =< 2 not constituting a safety risk based on investigator's judgment are acceptable
* Inadequately controlled hypertension (defined as systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg). Anti-hypertensive therapy to maintain a systolic blood pressure < 140 mmHg and/or diastolic blood pressure < 90 mmHg is permitted
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Patients with a baseline electrocardiography (EKG) demonstrating a QTc > 470 ms
* Serious non-healing or dehiscing wound, active ulcer or untreated bone fracture
* Proteinuria as demonstrated by urine dipstick or > 1 g of protein in a 24 hour urine collection. All patients with >= 2+ protein on dipstick urinalysis at baseline must undergo a 24 hour urine collection for protein
* Evidence of bleeding diathesis or clinically significant coagulopathy (in the absence of therapeutic anticoagulation)
* Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
* Subject with an uncontrolled seizure disorder, active neurologic disease, or active central nervous system (CNS) involvement except for individuals who have previously-treated CNS metastases, are asymptomatic, and have no requirement for doses of corticosteroids (indicated to reduce brain edema) higher than the equivalent of 10 mg of oral prednisone a day or anti-seizure medication for at least 2 weeks prior to first dose of study drug
* History of ongoing malignancies or malignancies in remission < 2 years. Adequately curative intent treated initial stage non-melanoma skin cancers; in situ carcinoma of the cervix; breast carcinoma in situ; low-grade local bladder cancer; and low-risk prostate cancer undergoing active surveillance will be allowed
* Pregnant women are excluded from this study. Based on its mechanism of action. Avelumab can cause fetal harm when administered to a pregnant woman. In animal models, the PD-1/PD-L1 signaling pathway is important in the maintenance of pregnancy through induction of maternal immune tolerance to fetal tissue. Human IgG1 immunoglobulins are known to cross the placenta. Therefore, avelumab has the potential to be transmitted from the mother to the developing fetus. Blockade of PD-L1 signaling has been shown in murine models of pregnancy to disrupt tolerance to the fetus and to result in an increase in fetal loss. Therefore, potential risks of administering avelumab during pregnancy include increased rates of abortion or stillbirth. Advise females of reproductive potential to use effective contraception during treatment with avelumab and for at least one month after the last dose of avelumab
* Lactating females: There is no information regarding the presence of avelumab in human milk, the effects on the breastfed infant, or the effects on milk production. Since many drugs including antibodies are excreted in human milk, advise a lactating woman not to breastfeed during treatment and for at least one month after the last dose of avelumab due to the potential for serious adverse reactions in breastfed infants
* Prior treatment with immune checkpoint inhibitor (e.g. anti-PD-1/PD-L1)
* Prior treatment with VEGF or VEGFR inhibitors (e.g. lenvatinib, bevacizumab)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renata Ferrarotto, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Ferrarotto R, Sousa LG, Feng L, Mott F, Blumenschein G, Altan M, Bell D, Bonini F, Li K, Marques-Piubelli ML, Dal Lago EA, Johnson JJ, Mitani Y, Godoy M, Lee A, Kupferman M, Hanna E, Glisson BS, Elamin Y, El-Naggar A. Phase II Clinical Trial of Axitinib and Avelumab in Patients With Recurrent/Metastatic Adenoid Cystic Carcinoma. J Clin Oncol. 2023 May 20;41(15):2843-2851. doi: 10.1200/JCO.22.02221. Epub 2023 Mar 10. PMID 36898078
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 participants enrolled from July 2019 to June 2021 (6 were screen failures).
Pre-assignment Details: Forty patients were enrolled from July 2019 to June 2021. Six were screen failures and thirty-four were treated.
Groups:
- Treatment (Axitinib, Avelumab): Axitinib was administered orally at 5 mg twice a day, and avelumab was administered intravenously at 10 mg/Kg on days 1 and 15 of 28-day cycles
Period: Overall Study
Arm/Group | Treatment (Axitinib, Avelumab)
Started | 34
Completed | 28
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Insurance Issues | 3
Not completed — Covid Restrictions | 2

BASELINE CHARACTERISTICS:
Population: 40 participants enrolled from July 2019 to June 2021 (6 were screen failures), 34 were treated and 6 of the 34 were evaluable for safety only and did not undergo the first re-staging imaging assessment
Arm/Group | Treatment (Axitinib, Avelumab)
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 7
Age, Continuous [Median (Full Range); unit: years] | 58 [29 to 88]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 34 were treated and 6 of the 34 were evaluable for safety only and did not undergo the first re-staging imaging assessmen
  Participants
    number analyzed (Participants) | 28
    Female | 16
    Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 34 were treated and 6 of the 34 were evaluable for safety only and did not undergo the first re-staging imaging assessmen
  Participants
    number analyzed (Participants) | 28
    Hispanic or Latino | 0
    Not Hispanic or Latino | 26
    Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 34 were treated and 6 of the 34 were evaluable for safety only and did not undergo the first re-staging imaging assessmen
  Participants
    number analyzed (Participants) | 28
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 7
    White | 16
    More than one race | 5
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Assess the Objective Response Rate (ORR) to Axitinib and Avelumab Combination According to RECIST 1.1 Criteria.
Description: All eligible patients who received at least one cycle of treatment and had at least one restaging image were considered evaluable for the primary end point. Objective response includes complete response (CR) + partial response (PR). Radiographic imaging for tumor assessment was performed at baseline and then every 8 weeks.
Time Frame: Up to 33 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Axitinib, Avelumab)
Number analyzed (Participants) | 28
percentage of participants | 18 [6.1 to 36.9]

2. Secondary Outcome: Estimate Median Progression-free Survival, Median Overall Survival
Description: Progression-free survival (PFS) was defined as the duration from start of treatment to date of progression or death, whichever occurred first. Overall survival (OS) was defined as the duration from start of treatment to death. The Kaplan-Meier approach was used to estimate the PFS and OS distributions, along with median estimates with 95% CI.
Time Frame: up to 40 months
Population: Forty patients enrolled from July 2019 to June 2021 (6 were screen failures), 34 were treated and 6 of the 34 were evaluable for safety only and did not undergo any re-staging imaging assessment, 28 were evaluable for time-to-event outcomes.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Axitinib, Avelumab)
Number analyzed (Participants) | 28
months
  PFS | 7.3 [3.7 to 11.2]
  OS | 16.6 [12.4 to NA] — Value not reached.

3. Secondary Outcome: Estimate Progression Free Survival Rate at 6 Months After Start of Treatment, Overall Survival Rate 6 Months After Start of Treatment
Description: Progression-free survival (PFS) was defined as the duration from start of treatment to date of progression or death, whichever occurred first. The PFS rate at 6-month was the percentage of patients without disease progression at 6 months. Overall survival (OS) was defined as the duration from start of treatment to death. The OS rate at 6-month was the percentage of living patients at 6 months. The Kaplan-Meier approach was used to estimate the PFS and OS distributions, along with median estimates with 95% CI.
Time Frame: completed at 6 months from start of treatment
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Axitinib, Avelumab)
Number analyzed (Participants) | 28
percentage of participants
  PFS rate at 6-month | 57 [41.5 to 78.8]
  OS rate at 6-month | 86 [73.7 to 99.7]

4. Secondary Outcome: Estimate Duration of Response
Description: Duration of response (DoR) was measured from the date response criteria were met until the first date that progression was documented. The Kaplan-Meier approach was used to estimate the DOR distributions, along with median estimates with 95% CI.
Time Frame: Up to 30 months
Population: Forty patients enrolled from July 2019 to June 2021 (6 were screen failures), 34 were treated and 6 of the 34 were evaluable for safety only and did not undergo any re-staging imaging assessment, 28 were evaluable for objective response and time-to-event outcomes. Five patients achieved confirmed partial response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Axitinib, Avelumab)
Number analyzed (Participants) | 5
months | 11 [5.5 to NA] — Value not reached.

5. Secondary Outcome: Evaluate Safety and Toxicity
Description: Evaluated for the number of incidences for safety and toxicity for treatment related adverse events that occurred in > 10% of patients and all grade 3 or higher treatment related adverse events.
Time Frame: Up to 30 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Axitinib, Avelumab)
Number analyzed (Participants) | 34
Participants
  Adverse Events | 34
  Serious Adverse Events | 7
  Labs | 19
  Deaths | 1

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed up to 30 months, All- Cause Mortality monitored/assessed up to 40 months. Adverse events were monitored until off study due to disease progression, death, unacceptable toxicity, consent withdrawal, or physician's discretion.
Description: All eligible participants who received at least one cycle of treatment were considered evaluable for safety analyses. AEs (related and unrelated) were graded according to Common Terminology Criteria for AEs version 4.0.
Arm/Group | Treatment (Axitinib, Avelumab)
All-Cause Mortality (participants affected / at risk) | 1/34
Serious Adverse Events (participants affected / at risk) | 7/34
Other Adverse Events (participants affected / at risk) | 31/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Axitinib, Avelumab) (N=34)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Transaminitis (Investigations) | 1 (1)
SOB (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
neoplasm pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Axitinib, Avelumab) (N=34)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 5 (8)
Alkaline phosphatase increased (Investigations) | 2 (3)
Allergic reaction (Investigations) | 2 (2)
Anemia (Investigations) | 4 (6)
Anorexia (Investigations) | 7 (8)
Anxiety (Investigations) | 1 (1)
Arthralgia (Investigations) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Blurred vision (Eye disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 3 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Creatinine increased (Investigations) | 3 (5)
Diarrhea (Gastrointestinal disorders) | 12 (21)
Dizziness (Nervous system disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysesthesia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Ear and labyrinth disorders - Other, specify (Earache B/L) (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Endocrine disorders - Other, specify (Low cortisol levels) (Endocrine disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Eye disorders - Other, specify (right eye fasciculations) (Eye disorders) | 1 (1)
Eye disorders - Other, specify (diplopia) (Eye disorders) | 1 (1)
Eye disorders - Other, specify (Left eye droop) (Eye disorders) | 1 (1)
Eye disorders - Other, specify (Loss of vision (both eyes)) (Eye disorders) | 1 (2)
Eye pain (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 22 (32)
Floaters (Vision floaters (left is greater than right)) (Eye disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Gait disturbance (General disorders) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (C. diff) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Epigastric) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastric pain) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (hematochezia) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Stomach infection) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (stomatitis) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Thick saliva) (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (Left leg weakness) (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (Asthenia) (General disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (5)
Hepatobiliary disorders - Other, specify (Deep Vein Thrombosis left arm) (Hepatobiliary disorders) | 1 (1)
HiccupsHiccups (Hepatobiliary disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Hypercalcemia (Metabolism and nutrition disorders) | 5 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypertension (Vascular disorders) | 10 (14)
Hypertension (Vascular disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Hypotension (Vascular disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 5 (5)
Infusion related reaction (General disorders) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Left ear bleeding (intermittent)) (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Investigations - Other, specify (Transaminitis) (Investigations) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 10 (10)
Musculoskeletal and connective tissue disorder - Other, specify (bilateral lower extremity muscle a (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Cramping hands and feet) (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Hip pain) (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Left shoulder blade) (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (leg pain) (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Muscle ache 4th-5th right rib) (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Shoulder Pain) (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Swollen left knuckle) (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Left shoulder pain) (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Abdominal pain) (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Nervous system disorders - Other, specify (Restless legs) (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, specify (neuropathic) (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Oral pain (Sore mouth) (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 (12)
Papulopustular rash (Infections and infestations) | 1 (1)
Paresthesia (Nervous system disorders) | 3 (3)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Portal vein thrombosis (deep vein thrombosis) (Hepatobiliary disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other, specify (Bronchitis) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Runny nose) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Sinus infection) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Itchy skin) (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Lip ulcer) (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Pruritic rash) (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Surgical and medical procedures - Other, specify (Colonoscopy) (Surgical and medical procedures) | 1 (1)
Surgical and medical procedures - Other, specify (Repair of reducible inguinal hernia) (Surgical and medical procedures) | 1 (1)
Surgical and medical procedures - Other, specify (Thoracentesis) (Surgical and medical procedures) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Uveitis (Eye disorders) | 1 (1)
Vascular disorders - Other, specify (Ecchymosis) (Vascular disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Weight loss (Investigations) | 9 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/71/NCT03990571/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/71/NCT03990571/ICF_001.pdf